CLINICAL TRIAL: NCT02231567
Title: Effectiveness of Neurocognitive Rehabilitation in Pain Management and Functional Recovery After Hip Replacement: Randomized Controlled Trial
Brief Title: Neurocognitive Rehabilitation After Hip Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, medical director, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3298/2014
Record Dates: First submitted 2014-08-08; First posted 2014-09-04 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2016-01

CONDITIONS: Hip Osteoarthritis
Keywords: hip replacement; neurocognitive rehabilitation; WOMAC questionnaire
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neurocognitive Rehabilitation (Experimental): Rehabilitative approach based on exercises proposed as sensory-motor problems, whose solution involves the use of higher cognitive functions (attention, memory, language).
  Interventions: Other: Neurocognitive Rehabilitation
- Traditional Rehabilitation (Active Comparator): It is a rehabilitative approach based on exercises for the recovery of hip's range of motion, muscle strengthening exercises, stretching exercises of the hamstring muscles, adductor and iliopsoas and proprioceptive exercises.
  Interventions: Other: Traditional Rehabilitation

INTERVENTIONS:
Other: Neurocognitive Rehabilitation — The patients will be treated in inpatient clinic with a neurocognitive rehabilitation approach. The frequency will be two times a day for six days a week for four consecutive weeks. Followed by outpatient treatment three times a week for four weeks. Each session lasts about one hour.
  Arms: Neurocognitive Rehabilitation
Other: Traditional Rehabilitation — The patients will be treated in inpatient clinic with a traditional rehabilitation approach. The frequency will be two times a day for six days a week for four consecutive weeks. Followed by outpatient treatment three times a week for four weeks. Each session lasts about one hour.
  Arms: Traditional Rehabilitation

SUMMARY:
The purpose of the study is to evaluate the effectiveness of an approach based on neurocognitive rehabilitation exercises in the form of sensory-motor problems, whose solution involves the use of higher cognitive functions (attention, memory, language), not required in a traditional approach proprioceptive, in order to obtain a more complete and long-lasting recovery.

ELIGIBILITY:
Inclusion Criteria:

* Presence of symptomatic unilateral primary hip osteoarthritis treated with surgical replacement with a posterior-lateral approach and the use of a non-cemented prosthesis (press-fit). All the implants are composed of a stem Symax (Stryker-Howmedica) and a ceramic head with coupling ceramic-ceramic and are implanted by the same surgeon.

Exclusion Criteria:

* Different diagnosis from hip osteoarthritis (eg. Fracture)
* Concomitant osteoarthrosis of the hip or knee with gait restrictions
* Lameness for more than six months
* Central nervous system or Peripheral nervous system disorders
* Systemic inflammatory disorders (eg. Rheumatoid Arthritis)
* Systemic infectious disorders
* Cognitive impairment
* Neoplastic disorders
* Surgical revisions
* Intraoperative complications
* Suspected hip replacement infection
* Hip replacement with endoprosthesis.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change of WOMAC Questionnaire from baseline to 24 weeks | baseline, 1 week, 8 weeks, 16 weeks, 24 weeks
  Questionnaire for the assessment of pain, stiffness and physical function. It measures physical function and symptoms of the lower limb and explores the impact of disability and pain on activities of daily living. The questionnaire is self-administered and it is based on a metric scale ranging from 0 (no difficulty) to 100 (extreme difficulty).

SECONDARY OUTCOMES:
Change of Barthel Index from baseline to 24 weeks | baseline, 1 week, 8 weeks, 16 weeks, 24 weeks
  Index for the evaluation of patient's performance in activities of daily living. The index is divided into eleven sub-categories that assess activities of daily living (ability to feed themselves, to ensure personal hygiene and dressing) and the mobility of the individual (gait, postural changes and transfers, stairs). For each item is assigned a score variable from full to reduced or absent functionality. The questionnaire is administered by an examiner and is based on a metric scale ranging from 0 (total dependence) to 100 (minimum dependence).
Change of Visual Analogue Scale (VAS) from baseline to 24 weeks | baseline, 1 week, 8 weeks, 16 weeks, 24 weeks
  It is based on a ten point scale, where 0 means no pain and 10 means the greatest pain ever. It enables the patients to express their pain intensity as numerical value.
Change of SF-36 Health Survey Questionnaire from baseline to 24 weeks | baseline, 1 week, 8 weeks, 16 weeks, 24 weeks
  Assessment of health status using the SF-36 Health Survey Questionnaire. The questionnaire is divided into eight sub-categories that measure the physical activity, role limitations due to physical health and emotional problems, physical pain, the perception of general health, vitality, social activities, mental health and changes in health status and two indices that summarize the overall assessment of the subject with respect to his physical health (ISF) and mental (ISM). Indices are derived from 8 subcategories evaluated and allow to summarize the results. The questionnaire is self-administered and subcategories is that the indices are based on a metric scale ranging from 0 (worst health status) to 100 (best health status) 17, 18.
Change of Psychological Well-Being Questionnaire (PWB) from baseline to 24 weeks | baseline, 1 week, 8 weeks, 16 weeks, 24 weeks
  Questionnaire for the assessment of psychological well-being and positive functioning of the individual. It includes 84 items and measures the six dimensions /scales of well-being proposed in the model developed by the American psychologist Carol Ryff: self-acceptance, positive interpersonal relationships, autonomy, environmental control, personal growth and purpose in life. The questionnaire is self-administered and each item is evaluated by a metric scale ranging from 1 (disagree) to 6 (totally agree). The negatively worded items are counted in reverse order. The sum score for each scale is calculated by summing the degree of agreement of each item.
Change of parameters of Gait Analysis from baseline to 24 weeks | baseline, 1 week, 8 weeks, 16 weeks, 24 weeks
  It's used to define the pattern of gait. The Gait Analysis provides different types of information such as quantitative kinematics data (angles of flexion-extension, abduction-adduction and external rotation of the main joints), velocity data (moments and powers the major joints) and electromyographic data.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Maria Saraceni, Principal Investigator — Umberto I Hospital, Sapienza University of Rome
Locations (1):
- Umberto I Hospital, Rome, Italy